CLINICAL TRIAL: NCT02693366
Title: Safety Study of the Endovascular Infusion of Bone Marrow Derived Mononuclear Cells in Patients With Focal Segmental Glomerulosclerosis
Brief Title: Stem Cell Therapy for Patients With Focal Segmental Glomerulosclerosis
Acronym: STEFOG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other); Ministry of Health, Brazil (Other Government); National Research Council, Brazil (Other); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Marcelo Marcos Morales, MD, PhD, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE:01498412.5.0000.5257
Record Dates: First submitted 2016-01-30; First posted 2016-02-26 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Focal Segmental Glomerulosclerosis; Chronic Kidney Diseases
Keywords: bone marrow cells; Focal Segmental Glomerulosclerosis; Chronic Kidney Diseases; stem cell; cell therapy
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Renal Insufficiency, Chronic | interventions — Bone Marrow Purging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Cell Therapy (Experimental): We are conducting a prospective, non-randomized, single-center longitudinal study in five patients with progressive chronic kidney disease and estimated clearance between 40 and 20 ml / min. Patients will be followed by clinical and laboratory examination for 3 months prior to the procedure. These previous results serve as a control for comparison with a second time when the same patients receive treatment with stem cells being subsequently followed up for 9 months a total of one year of clinical follow-up.
  Interventions: Other: Bone marrow stem cell

INTERVENTIONS:
Other: Bone marrow stem cell — Endovascular infusion of bone marrow derived cells in both renal arteries.

SUMMARY:
The purpose of this study is to analyze the safety, renal function, metabolic disorders and quality of life data in patients with focal segmental glomerulosclerosis treated with endovascular infusion of bone marrow derived mononuclear cells.

DETAILED DESCRIPTION:
Will be studied five patients with progressive chronic kidney disease and estimated clearance between 40 and 20 ml / min. Patients will be followed by clinical and laboratory examination for 3 months prior to the procedure. These previous results serve as a control for comparison with a second time when the same patients receive treatment with stem cells being subsequently followed up for 9 months a total of one year of clinical follow-up.

Bone marrow aspiration and subsequent cell preparation were accomplished on the same day as the endovascular infusion of autologous Bone Marrow derived Mononuclear stem cells (BMDMCs) in both renal arteries. Collection was performed under spinal anesthesia and light sedation, through puncture and repeated aspirations at the posterior iliac crest region. A total of 80 mL of bone marrow aspirate was collected from each patient, and after removal of bone and fatty residues, mononuclear cells were isolated by a Ficoll-Paque Plus (Amersham Biosciences, São Paulo, Brazil).For each patient, 2×107 cells will be labeled with 99mTc. Briefly, 500 μl of sterile SnCl2 solution is added to the cells and the mixture is incubated at room temperature for 10 min. Forty-five millicurie (mCi) of 99mTc is then added and incubation continued for another 10 min. After centrifugation (500×g for 5 min), the supernatant is removed and the cells are washed in saline solution. The pellet will be also resuspended in saline solution. Viability of the labeled cells will be assessed by the trypan blue exclusion test, and estimated to be greater than 93% in all cases.The labeling efficiency (%) will be calculated by the activity in the pellet divided by the sum of the radioactivity in the pellet plus supernatant and estimated to be greater than 90% in all cases.

After the collection of the stem cells, the patient will be submitted to puncture the femoral artery using the Seldinger technique under local anesthesia, followed by catheterization of the ostium of the renal arteries with minimum use of nonionic iodinated contrast. With the routing of diagnostic catheter or guide, the solution numbering about 30 to 100 million of dissolved plasma cells will be divided and injected into two renal arteries. The infusion volume is about 5 ml in each kidney. Whole body and planar scans will be performed 2 and 24h after infusion to determine the migration and cell viability. The patient will remain hospitalized for more 48 hours for clinical monitoring and collection of laboratorial tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of primary focal segmental glomerulosclerosis after having been previously treated with corticosteroids and immunosuppressive drugs and have not reached satisfactory answer. Will also be considered candidates those patients who performed late diagnosis and therefore no more clinical indication to perform therapy with corticosteroids and immunosuppressants. In both cases, showing irreversible loss of renal function with filtration rate between 40 - 20 ml/min.
* Patient should use the classical nephroprotective medication: angiotensin-converting enzyme inhibitor or angiotensin-receptor blocker, or both.

Exclusion Criteria:

* Acute urinary tract infection;
* Urinary infection with tuberculosis bacillus or fungi;
* Patients with poorly anatomical formations of the urinary tract, polycystic kidney disease and other congenital or acquired kidney diseases.
* Blood pressure greater than 160 mm Hg systolic and 100 mmHg diastolic, in measurements taken during the last 3 outpatient visits;
* Who has performed examination with iodinated contrast the last 3 months
* Use of potentially nephrotoxic drugs;
* Use of corticosteroid therapy in immunosuppressive doses or more than 0.3 mg/kg/day
* Inability to obtain vascular access for endovascular procedure
* Sepsis (defined according to the Society of Critical Care Medicine, American College of Chest Physicians, 1992);
* Malignancies
* Autoimmune disorders,
* Neurodegenerative diseases;
* Acute heart failure or decompensated;
* Primary hematologic diseases;
* Osteopathies reflecting increased risk for spinal puncture;
* Coagulopathies;
* Liver failure;
* History of stroke or myocardial infarction in the last 6 months;
* Pregnancy or breastfeeding;
* History and serology of chronic infectious diseases, including HIV, Hepatitis C virus, Hepatitis B virus
* Participation in another clinical trial last year
* Cognitive impairment to understand all procedures
* Prolonged travel plans or domicile changes to other states that generate unable to attend the follow-up visits;
* Any other clinically significant active disease in the opinion of the principal investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-06-25 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Kidney injury | 9 months
  Increase of serum creatinine of about 0.5 mg / dL when levels are less than 3.0 mg / dl and 1.0 mg / dl baseline levels when are greater than or equal to 3.0 mg / dL) when confirmed with the second examination.
  * Acute: evaluated within 15 days of cell therapy;
  * Subacute: evaluated 15-90 days of cell therapy
Chronic kidney disease | 9 months
  Doubling of serum creatinine based on the third month after the cell therapy or the need to start dialysis
Potential differentiation disorders of transplanted cells | 9 months
  Analyzed by clinical and imaging tests such abdominal ultrasound and chest radiography
Systemic inflammatory potential of mononuclear cells administration in renal circulation | 9 months
  Laboratory tests: C-reactive protein, erythrocyte sedimentation rate, blood count and urinary sediment
Death | 9 months

SECONDARY OUTCOMES:
Renal function | 9 months
  The estimated creatinine clearance assessment by MDRD formula
Bone metabolism | 9 months
  Evaluation of bone metabolism by serum phosphorus (mg/dL), calcium (mg/dL), parathormone (pg/ml), 25 (OH) vit. D (ng/ml).
Balance assessment electrolyte and acid-base | 9 months
  Balance assessment electrolyte and acid-base by serum sodium (mEq/l), potassium (mEq/l), uric acid (mg/dl) and bicarbonate
The lipid profile assessment and anemia | 9 months
  The lipid profile assessment (LDL- cholesterol, HDL-cholesterol and triglyceride) and anemia measured by hemoglobin (g/dL) and hematocrit.
Quality of life questionnaire | 9 months
  Clinical improvement of the patient, with subjective assessment of general health and well being through SF36 quality of life questionnaire
Imaging tests | 9 months
  Imaging tests: Renal scintigraphy with 99mTc-DTPA and DMSA

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Marcos Morales, MD,PHD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universitary Hospital Clementino Fraga Filho - UFRJ, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Botelho BF, Barreira AL, Filippo MG, Asensi KD, Faccioli LAP, Dos Santos Salgado AB, de Salles EF, Marques CEC, Silva PL, Dos Santos Goldenberg RC, Maiolino A, Gutfilen B, de Souza SAL, Junior ML, Morales MM. Safety and Biodistribution of an Autologous Bone Marrow-Derived Mononuclear Cell Infusion into Renal Arteries in Patients with Focal Segmental Glomerulosclerosis: A Phase 1 Study. Stem Cells Int. 2024 Jul 9;2024:2385568. doi: 10.1155/2024/2385568. eCollection 2024. PMID 39015674